CLINICAL TRIAL: NCT04469010
Title: Efficacy Evaluation of 16 Weeks' Dietary Supplementation With Iron Bis-glycinate Plus Vitamin C on Cognitive Function, Subjective Mood, Fatigue, Health and Well-being in Non-anaemic Iron Deficient and Iron Sufficient Women of Reproductive Age
Brief Title: Efficacy Evaluation of 16 Weeks' Dietary Supplementation With Iron Bis-glycinate Plus Vitamin C on Cognitive Function, Subjective Mood, Fatigue, Health and Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 9BN1
Record Dates: First submitted 2020-07-09; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2019-07

CONDITIONS: Cognitive Function and Mood; Non-anaemic Iron Deficiency
Keywords: Cognition; Mood; Fatigue; Well-being; Women's health; Iron supplementation; Vitamin C
MeSH Terms: conditions — Fatigue | interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Participants will receive either iron and vitamin C, iron alone or placebo for a period of 16 weeks to consume daily
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Iron and Vitamin C (Experimental): 28mg iron bis-glycinate chelate and 240mg vitamin C
  Interventions: Dietary Supplement: Iron Bis-Glycinate Chelate and Vitamin C
- Iron (Active Comparator): 28mg iron bis-glycinate chelate
  Interventions: Dietary Supplement: Iron Bis-Glycinate Chelate
- Placebo (Placebo Comparator): Matched placebo tablets
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Iron Bis-Glycinate Chelate and Vitamin C — 28 mg iron 240 mg vitamin C
  Arms: Iron and Vitamin C
Dietary Supplement: Iron Bis-Glycinate Chelate — 28 mg iron
  Arms: Iron
Dietary Supplement: Placebo — Matched placebo
  Arms: Placebo

SUMMARY:
Iron deficiency is the most prevalent nutritional deficiency worldwide with one in four estimated to be affected by iron deficiency anaemia. Women of reproductive age are at greatest risk for iron deficiency and anaemia due to iron losses during menstruation and childbirth as well as the increased need for iron throughout pregnancy. However, iron deficiency without anaemia is at least twice as common as iron deficiency anaemia with females aged 11-49 at the biggest risk of all. Despite this, it is commonly left undiagnosed. Those who are iron deficient non-anaemic can still suffer from the same common consequences of iron deficiency anaemia; these include unexplained fatigue, mood changes and decreased cognitive performance. However, randomised controlled trials (RCTs) assessing the effect of iron supplementation upon cognitive performance, mood, fatigue and well-being in non-anaemic iron deficient women of reproductive age are limited. There is also a lack of well-defined diagnostic criteria for non-anaemic iron deficiency, which makes comparisons across RCTs difficult. However, there is evidence to suggest that a haemoglobin cut off of ≥120 g/L and serum ferritin ≤ 20 µg/L provides an accurate indication of non-anaemic iron deficiency in women of reproductive age; this is inclusive of the ability to recognise iron-associated deficits in psychological and physiological functioning. Additionally, previous RCTs could be improved by utilising a lower dose of iron in a bis-glycinate chelate form, which is evidenced to have superior bioavailability, tolerability and subsequent efficacy compared to ferrous formulations. Iron bis-glycinate absorption is also negatively associated to serum ferritin levels, which is suggestive of a non-anaemic iron deficient population benefitting most from it's administration. The current study aims to build upon previous iron RCTs in populations of non-anaemic iron deficient and iron sufficient women of reproductive age by investigating the effects of 16-weeks supplementation with either iron bis-glycinate chelate alone, iron bis-glycinate plus vitamin C (as ascorbic acid) or matched placebo upon cognitive performance, subjective mood, fatigue, health and well-being.

DETAILED DESCRIPTION:
Each participant will be required to attend the laboratory on four occasions. The first is comprised of a screening/training visit, which will take place in the afternoon for approximately 2.5 hours. This will also be between days 21-28/ the week before onset of their menstrual cycle. If they do not have menstrual bleeds then this appointment can be any afternoon. This will comprise: briefing of requirements of the study; obtaining of informed consent; confirmation of eligibility to take part, including collection of demographic data and health screening, and training on the cognitive and mood measures. The training session will follow standard operating procedures to decrease the chance of learning effects during main trials. Extra training will be given where necessary.

Participants will be required to complete questionnaires based upon food frequency, caffeine consumption and to estimate the number of hours of exercise completed on a weekly basis. A menstrual cycle questionnaire will also be completed to estimate menstrual blood loss and so that participants attend their testing visit during days 7-14 of their cycle. If participants do not have a menstrual cycle due to contraceptive methods, then appointments will be approximately two weeks apart. A finger-prick and venous blood sample will be collected from participants, which will be analysed for iron status. Those whose haemoglobin levels are <120g/L will be advised to seek advice from their GP. Participants who fell into the iron status category of iron sufficient (haemoglobin ≥120 g/L and serum ferritin > 20 µg/L) or non-anaemic iron deficient (haemoglobin ≥120 g/L and serum ferritin ≤ 20 µg/L) will be informed of their eligibility for the intervention study by email or phone between the initial visit and their next.

For the testing visit, participants will be asked to fast for 12 hours prior to the visit, avoiding intake of all food and drink with the exception of water. They will also be asked to avoid alcohol and refrain from intake of 'over the counter' medication for 24 hours. Participants will arrive at the laboratory at a designated time in the morning. The following procedures will take place prior to cognitive and mood testing:

* Review of continued conformity to eligibility criteria
* Adverse event and concomitant medication assessment
* Ensure that participant is in good health Participants will then complete the baseline cognitive and mood assessments. Following this, participants are informed of their iron status and will be briefed regarding the requirements of the intervention study. Following this, informed consent will be obtained prior to randomising participants to one of three treatments and providing them with a treatment diary to log treatment consumption and any adverse events experienced.

Participants will return to the laboratory after 8 weeks to exchange treatment bottles and diaries in order to check compliance.

Participants will finally return to the laboratory after a further 8 weeks (16 weeks total). The same procedures will take place prior to cognitive and mood testing as completed at the baseline testing visit, with the addition of finger prick and venous blood sample and weight measurement. Participants will then complete the same cognitive and mood assessments as completed during the baseline testing visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Female
* Aged 18-49 (inclusive)
* Have a BMI of between 18.5-40
* Have an English bank account (required for payment)

Exclusion Criteria:

* Aged under 18 or above 49 years
* BMI lower than 18.5 or higher than 40
* Pre-existing medical condition/illness with some exceptions - please check with researcher
* Blood disorders (including anaemia) or any known active infections
* Current or past breast cancer diagnosis and/or mastectomy
* Smoking or use of any nicotine replacement products e.g. vaping, gum, patches
* Pregnant, trying to get pregnant or breast feeding
* Currently taking any prescription medication with some exceptions - please check with researcher
* Food allergies/sensitivities relevant to the study
* Regular use of dietary/herbal supplements within the last month (defined as more than 3 consecutive days or 4 days in total)
* Use of iron supplements within the past 4 months
* Have donated more than 300ml of blood in the past 3 months
* Have haemoglobin levels below 120g/L
* History of significant head trauma or suffer from frequent migraines that require medication (more than or equal to one per month)
* Learning difficulties, dyslexia, or colour blindness
* Visual impairment that cannot be corrected with glasses or contact lenses
* Currently taking part in any other clinical or nutritional intervention studies or have in the past 4 weeks
* Any health condition that would prevent fulfillment of the study requirements

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants must be female as assigned at birth
Enrollment: 151 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
Speed of attention | 16 weeks
  An overall score for Speed of attention will be derived by calculating the average score from 3 separate standardised task outcomes (ZChoice reaction time correct reaction time + ZRapid visual information processing correct reaction time + ZDigit vigilance correct reaction time) /3
Subjective fatigue | 16 weeks
  Subjective fatigue will be derived from the total score of the Piper Fatigue Scale. Scores range from 1 to 10. Higher scores are indicative of greater fatigue.

SECONDARY OUTCOMES:
Accuracy of episodic memory | 16 weeks
  An overall score for episodic memory will be derived by calculating the average score from 4 separate standardised task outcomes (Zimmediate word recall accuracy + Zdelayed word recall accuracy + Zword recognition accuracy + Zpicture recognition accuracy)/4
Speed of episodic memory | 16 weeks
  An overall score for speed of memory will be derived by calculating the average score from 2 separate standardised task outcomes (Zpicture recognition correct reaction time + Zword recognition correct reaction time)/2
Accuracy of attention | 16 weeks
  An overall score for accuracy of attention will be derived by calculating the average score from 3 separate standardised task outcomes (ZChoice reaction time accuracy + ZZRapid visual information processing accuracy + ZZDigit Vigilance accuracy)/3
Accuracy of executive function | 16 weeks
  An overall score for executive function will be derived by calculating the average score from 5 separate standardised task outcomes (Znumeric working memory accuracy + ZZserial 3 subtractions accuracy + ZZserial 7 subtractions accuracy + ZStroop accuracy - ZPeg and Ball errors)/5
Speed of executive function | 16 weeks
  An overall score for speed of executive function will be derived by calculating the average score from 3 separate standardised task outcomes (Znumeric working memory correct reaction time + Zstroop correct reaction time + ZPeg and Ball overall reaction time)/3
Computerised location learning task | 16 weeks
  An overall score is calculated utilising the total displacement over the 5 learning trials to create a total learning index score. Scores range from 0 to 1.
Subjective overall mood disturbance | 16 weeks
  Subjective mood disturbance is derived from the overall score of the Profile of Mood States questionnaire. Higher scores indicate a greater degree of overall mood disturbance.
Subjective sleep quality | 16 weeks
  Subjective sleep quality is derived from the overall score of the Sleep Condition Indicator. Total scores ranged from 0 to 32. Higher scores are indicative of greater subjective sleep quality.
Subjective stress | 16 weeks
  Subjective stress is derived from the overall score of the Perceived Stress Scale. Higher scores are indicative of greater subjective stress
Health outcomes | 16 weeks
  Subjective health outcomes are derived from the SF-12. Scores range from 0 to 100. Higher scores are indicative of better self-reported health.
Subjective alertness | 16 weeks
  Subjective alertness will be derived from an Alertness visual analogue scale presented following cognitive task performance. Scores range from 0 to 100. Higher scores are indicative of greater feelings of alertness.
Subjective mental fatigue | 16 weeks
  Subjective mental fatigue will be derived from a Mental Fatigue visual analogue scale presented following cognitive task performance. Scores range from 0 to 100. Higher scores are indicative of greater feelings of mental fatigue.
Global accuracy | 16 weeks
  An overall score for global accuracy will be derived by calculating the average score from 13 separate standardised outcomes (ZChoice reaction time accuracy + ZZRapid visual information processing accuracy + ZNumeric working memory accuracy + ZZDigit Vigilance accuracy + ZStroop accuracy - ZPeg and Ball Errors + ZZSerial 3 subtractions accuracy + ZZSSerial 7 subtractions accuracy + ZPicture recognition accuracy + ZWord recognition accuracy + ZImmediate word recall accuracy + ZDelayed word recall accuracy + ZZComputerised location learning accuracy)/13
Global speed | 16 weeks
  An overall score for global speed will be derived by calculating the average score from 8 separate standardised outcomes (ZChoice reaction time correct reaction time + ZNumeric working memory correct reaction time + ZDigit vigilance correct reaction time + ZZPeg and Ball overall reaction time + ZStroop correct reaction time + ZPicture recognition correct reaction time + ZWord recognition correct reaction time + ZRapid visual information correct reaction time) /8

CONTACTS AND LOCATIONS:
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom